CLINICAL TRIAL: NCT00119782
Title: Reducing Obesity at the Workplace: a Randomized Trial
Brief Title: Promoting Activity and Changes in Eating (PACE) to Reduce Obesity
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Shirley A. A. Beresford, PhD, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 193; R01HL079491 (NIH)
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Obesity; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Heart Diseases | interventions — Diet; Exercise; Environment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Comprehensive worksite intervention
  Interventions: Behavioral: Diet; Behavioral: Exercise; Behavioral: Environment
- 2 (Experimental): Delayed intervention control group
  Interventions: Behavioral: Diet; Behavioral: Exercise; Behavioral: Environment

INTERVENTIONS:
Behavioral: Diet — A dietary intervention that will promote lower calorie intake
Behavioral: Exercise — A physical activity intervention combining increased daily physical activity and regular, structured exercise
Behavioral: Environment — Increase worksite access to both healthy foods and physical activity

SUMMARY:
Reducing the prevalence of obesity in the population is one of the Healthy People 2010 goals. Increased vigilance is required in all age groups in preventing and reversing overweight and obesity. On an individual level, behavioral factors that influence body weight include eating choices leading to excess calorie intake and physical activity patterns leading to diminished calorie expenditure. An imbalance between the two over time leads to increased weight. On a population basis, the prevalence of overweight is associated with a myriad of influences, including social, behavioral, cultural, and environmental factors as well as genetic and physiological factors. For a majority of overweight individuals, restoring a balance between energy intake and expenditure is difficult, and therefore there is an increasing emphasis on preventing obesity on a population level. The long-term goal of this research is to prevent further increase in rates of obesity in the population. In the adult population of working age, a majority of the day is spent in the worksite, suggesting that interventions at the worksite level may offer the opportunity for success in this age group. It is anticipated that this project will yield important contributions to the understanding of obesity prevention.

DETAILED DESCRIPTION:
BACKGROUND:

More than half of American adults are overweight or obese, and this proportion is increasing. The health risks associated with obesity include diabetes, cardiovascular disease, arthritis, and some cancers. It is well established that on an individual level, weight gain is caused by taking in more calories than are expended. On a population basis, the prevalence of overweight and obesity is associated with a myriad of influences, including genetic and physiological factors as well as social, behavioral, cultural, and environmental factors. Behavioral factors that contribute to weight gain include eating choices that lead to increased energy intake and physical activity choices that lead to decreased energy expenditure. For a majority of overweight individuals, restoring the balance between energy intake and expenditure is difficult.

DESIGN NARRATIVE:

This study will develop and test a comprehensive intervention involving simple messages that will integrate changes in dietary intake with changes in energy expenditure, while simultaneously modifying structural and environmental factors to promote social support and opportunities for behavioral change. The study will recruit and randomize 48 worksites to a 2-year intervention in which the following will be carried out: build a physical activity intervention combining increased daily physical activity and regular, structured exercise; build a dietary intervention that will promote lower calorie intake; and increase worksite access to both healthy foods and physical activity. The primary aim is to evaluate the effectiveness of the intervention in reducing or maintaining body mass index in a randomized controlled trial of worksites. The study will compare changes in body mass index in intervention versus control worksites using two cross-sectional surveys at baseline and follow-up. Additional assessments using biomarkers and fitness measures will be performed in a subset of employees. The research team has considerable experience with interventions at the worksite level and substantial expertise in obesity prevention.

ELIGIBILITY:
The study is enrolling employees only at participating worksites.

INCLUSION CRITERIA FOR WORK SITES:

* Meets specific standard industrial codes
* At least 20% of employees are sedentary
* Willing to provide a list of employees
* Able to achieve at least a 70% response rate to the baseline survey

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Body mass index | Measured at Month 24 follow-up visit; adjusted for baseline body mass index

SECONDARY OUTCOMES:
Self-reported dietary and physical activity behaviors | Measured at Month 24 follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Beresford, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States